CLINICAL TRIAL: NCT01858818
Title: Project 4: Acute Effects of Alcohol on Learning and Habitization in Healthy Young Adults
Acronym: LeAD_P4
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: ZI 1119/4-1
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Alcoholism
Keywords: CAIS Computer Assisted Infusion System; real life drinking behavior; family history of alcoholism; conditioning; instrumental learning; habitization
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy 18 year old males

SUMMARY:
This project aims to investigate how dysfunctional learning and habitization are affected by acute alcohol exposure, and whether individual differences in such alcohol effects can predict later development of Alcohol Use Disorders (AUDs). Eighty 18-year-old healthy male subjects are tested on two days in a within-subjects design with blinded administration of alcohol vs. placebo and different behavioral and learning tasks. The investigators investigate how alcohol influences the performance during these tasks, whether alcohol effects differ between high- and low-risk subjects, and whether task performance under alcohol predicts future AUDs.

DETAILED DESCRIPTION:
This project is part of a large multi-center study in Dresden and Berlin on Learning and Alcohol Dependence (LeAD). Project 4 aims to investigate how dysfunctional learning and habitization are affected by acute alcohol exposure, and whether individual differences in such alcohol effects can predict later development of AUDs. The project investigates eighty 18-year-old healthy male subjects, a subsample of LeAD project 1 that were already tested in Dresden using fMRI(Clinical Trials.govID: NCT01744834). Participants are tested on two days in a within-subjects design with blinded administration of alcohol or placebo. On 2 days participants are performing three behavioral and learning tasks measuring: 1. conditioning of money vs. drink stimuli 2. habitization vs. instrumental learning and 3. approach and avoidance behavior towards money and drink stimuli. The investigators investigate how alcohol influences the performance during these tasks, whether alcohol effects differ between high- and low-risk subjects, and whether task performance under alcohol predicts future AUDs. Participants will be followed up after three years. The project investigates whether single doses of alcohol affect the conditioning of monetary reward or alcoholic stimuli, impair instrumental learning, and enhance stimulus-response associations. The investigators want to test whether individual performance parameters are related to other risk factors for AUDs, e.g. family history of alcoholism or impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* men at age 18
* signed informed consent
* social drinking in the three months before participation participation, defined by at least two drinking days in any four weeks-interval
* ability to provide AUD information about biological parents and grandparents

Exclusion Criteria:

* lifetime history of Diagnostic Statistical Manual-IV bipolar or psychotic disorder
* current diagnosis of one of the following disorders: major depressive disorder, generalized anxiety disorder, PTSD, borderline personality disorder, or obsessive-compulsive disorder
* prior treatment for any axis-I or axis-II disorder except for specific disorders of childhood and adolescence (i.e., oppositional defiant disorder, conduct disorder, ADHD)
* history of substance dependence other than nicotine dependence
* current substance use other than nicotine and alcohol as evinced by positive urine screen
* history of severe head trauma or other severe central neurological disorder (e.g. multiple sclerosis)
* alcohol intake in the last 24 hours before test days
* use of medications or drugs known to interact with the central nervous system within the last 10 days or at least four half-lives post last intake

Ages: 18 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: random sampling of representative sample of 18 year old men in the area of Dresden
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
individual learning parameters | 2 days at age 18
  estimated by computational modeling of behavioral performance in learning/conditioning tasks the investigators test effects of individual parameters on actual risk factors of AUDs and future AUDs

SECONDARY OUTCOMES:
individual approach/avoidance reaction time differences | 2 days at age 18
  individual reaction time (RT) differences between approach and avoidance of alcoholic, non-alcoholic, and monetary stimuli under alcohol vs. placebo are measured the investigators test effects of individual RT differences on actual risk factors of AUDs and future AUDs

OTHER OUTCOMES:
lexical decision task performance | 2 days at age 18
  when deciding whether a word is a real word or not, accuracy should go down and reaction times up when people are alcoholized vs. sober the variable is used as a measure for general impairment of decision making and RT under alcohol

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Zimmermann, PD Dr., Principal Investigator — University Hospital Carl Gustav Carus at TU Dresden; Michael Smolka, Prof. Dr., Principal Investigator — Section of Systems Neuroscience at TU Dresden; Hans-Ulrich Wittchen, Prof. Dr., Study Chair — TU Dresden; Andreas Heinz, Prof. Dr., Study Chair — Charite University, Berlin, Germany
Locations (1):
- University Hospital Carl Gustav Carus, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Junger E, Javadi AH, Wiers CE, Sommer C, Garbusow M, Bernhardt N, Kuitunen-Paul S, Smolka MN, Zimmermann US. Acute alcohol effects on explicit and implicit motivation to drink alcohol in socially drinking adolescents. J Psychopharmacol. 2017 Jul;31(7):893-905. doi: 10.1177/0269881117691454. Epub 2017 Feb 21. PMID 28675116